CLINICAL TRIAL: NCT00765141
Title: A Multi-Center Protocol for Obtaining and Storing Human Samples for Immediate or Future Microbial, Immune, or Host Microbe Scientific Study
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled per PI discretion
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-011
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Infection
Keywords: wound debridement; removed orthopedic implants; removed catheters or shunts; excised tonsils; amputated tissue; sputum, stool; or other excretions.
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples can include material such as wound debridement, removed orthopedic implants, removed catheters or shunts, excised tonsils, amputated tissue, sputum, stool, or other excretions.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The intent of this protocol is to salvage human-related material that is normally destined for destruction, so it can be used in infection-related scientific studies.

DETAILED DESCRIPTION:
This clinical material can be studied in order to better understand the molecular, cellular, or ecological components of the infected or potentially infected tissue or device. These studies may be able to provide important insights into the keys of chronic infections, complex infections, medical biofilms, pathogen ecology, and healing.

ELIGIBILITY:
Inclusion Criteria:

* The Subject must be 18 years of age or older.
* The Subject must be mentally competent as determined by the Investigator.

Exclusion Criteria:

* The Subject may not be currently incarcerated.
* The Subject may not be knowingly pregnant.
* The Subject may not be institutionalized.
* The Subject may not be an employee or student of the investigator or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The samples can include material such as wound debridement, removed orthopedic implants, removed catheters or shunts, excised tonsils, amputated tissue, sputum, stool, or other excretions.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States